CLINICAL TRIAL: NCT02799173
Title: Determination of the RANKL/Osteoprotegerin Ratio in Patients With Systemic Lupus Erythematosus. Role in Osteoporosis and Cardiovascular Calcification
Acronym: CALCILUP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PHRCIR09-PR-MAZIERE-MME
Record Dates: First submitted 2016-06-10; First posted 2016-06-14 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Osteoporosis; Lupus Erythematosus, Systemic
Keywords: cardiovascular calcification; RANK: Receptor Activator of Nuclear Factor kappa B; RANKL: Receptor Activator of Nuclear Factor kappa B Ligand; OPG: Osteoprotegerin; SLE: Systemic lupus erythematosus
MeSH Terms: conditions — Osteoporosis; Lupus Erythematosus, Systemic | interventions — Ultrasonography, Doppler

ARMS (1):
- Systemic lupus erythematosus (Experimental): RANKL/OPG ratio bone densitometry fan beam CT scan Doppler ultrasound
  Interventions: Biological: RANKL/OPG ratio; Device: bone densitometry; Device: fan beam CT scan; Device: Doppler ultrasound

INTERVENTIONS:
Biological: RANKL/OPG ratio
Device: bone densitometry
Device: fan beam CT scan
Device: Doppler ultrasound

SUMMARY:
Patients with Systemic lupus erythematosus (SLE) are known to present an increased risk of osteoporosis and cardiovascular calcification. It has also been suggested that bone remodelling and cardiovascular calcification are regulated by the same mechanisms, but inversely in terms of calcium deposition, as osteoporosis is often associated with cardiovascular calcification. Inflammatory and immune factors have been implicated in these two processes.

The role of the RANKL/OPG system in osteoclast differentiation has been elucidated over the last ten years. RANKL induces differentiation of monocytes-macrophages into osteoclasts, while, inversely, OPG exerts an inhibitory role by inactivating RANKL. Differentiation of smooth muscle cells into osteoblasts in the vessel wall induces calcification, and this phenomenon is counterbalanced by differentiation of monocytes into osteoclasts. Although the role of the RANKL/OPG ratio in the pathogenesis of osteoporosis has now been clearly established, its role in vascular calcification is only hypothetical at the present time.

This study will focus on patients with SLE diagnosed and followed in the Amiens University Hospital Internal Medicine and Nephrology departments

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years old
* suffering from systemic lupus erythematosus.

Exclusion Criteria:

underlying diseases that can lead to bone and cardiovascular metabolic disturbances :

* Malignancies such as cancer metastasized
* Autoimmune disease other than LED or of overlap syndrome ( rhupus , MCTD )
* Infection by HIV, hepatitis B and C
* Hepatic Cirrhosis
* Chronic renal failure
* Parathyroid disorders

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2011-04-15 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

PRIMARY OUTCOMES:
RANKL/OPG ratio | Day 0
presence of osteoporosis | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Cécile MAZIERE, Md, PhD, Principal Investigator — CHU Amiens
Locations (2):
- France (2):
  - CHU Amiens, Amiens
  - CHU Rouen, Rouen